CLINICAL TRIAL: NCT00693420
Title: Safety and Efficacy of Bimatoprost Solution in Increasing Overall Eyelash Prominence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-032
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Results first posted 2009-05-12 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Eyelashes
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Bimatoprost 0.03% solution
  Interventions: Drug: Bimatoprost 0.03% sterile solution
- 2 (Placebo Comparator): Vehicle solution
  Interventions: Drug: vehicle sterile solution

INTERVENTIONS:
Drug: Bimatoprost 0.03% sterile solution — Apply one drop of study medication using single-use per eye applicator to upper eyelid margin once daily.
  Other Names: LUMIGAN®
  Arms: 1
Drug: vehicle sterile solution — Apply one drop of study medication using single-use per eye applicator to upper eyelid margin once daily
  Arms: 2

SUMMARY:
This study evaluates the safety and effectiveness of topical bimatoprost solution for enhancing eyelash prominence.

ELIGIBILITY:
Inclusion Criteria:

* Dissatisfaction with eyelash prominence,
* Eyelash prominence assessment of minimal or moderate,
* Ability to provide written informed consent

Exclusion Criteria:

* Subjects without visible lashes,
* Asymmetrical (uneven lashes or longer on one side than the other) eyelashes,
* Any eye disease or abnormality,
* Eye surgery,
* Permanent eyeliner,
* Eyelash implants,
* Eyelash extension application,
* Any use of eyelash growth products within 6 months of study entry,
* Treatments that may effect hair growth,
* Subjects requiring eye drop medications for glaucoma,
* Subjects having a situation or condition, which the study doctor feels might put you at risk, may make the study results confusing, or may interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- San Diego, California, United States
- Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Fagien S, Walt JG, Carruthers J, Cox SE, Wirta D, Weng E, Beddingfield FC 3rd. Patient-reported outcomes of bimatoprost for eyelash growth: results from a randomized, double-masked, vehicle-controlled, parallel-group study. Aesthet Surg J. 2013 Aug 1;33(6):789-98. doi: 10.1177/1090820X13495887. Epub 2013 Jul 19. PMID 23873891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Started | 137 | 141
Completed | 131 | 126
Not Completed | 6 | 15
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Sponsor Request - Conflict of Interest | 0 | 2
Not completed — Personal Reasons | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution | Total
Number analyzed (Participants) | 137 | 141 | 278
Age, Customized [Number; unit: participants]
  <45 years | 44 | 43 | 87
  Between 45 and 65 years | 82 | 88 | 170
  >65 years | 11 | 10 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 136 | 270
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least a 1-grade Increase on the Global Eyelash Assessment (GEA) Scale From Baseline to Week 16
Description: The GEA scale is an investigator-graded 4-point ordinal scale of overall eyelash prominence (1 [minimal], 2 [moderate], 3 [marked], 4 [very marked])
Time Frame: Baseline to Week 16
Population: Intent to Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
Percentage of participants
  Week 1 | 5.1 | 2.1
  Week 4 | 14.6 | 7.8
  Week 8 | 50.4 | 14.9
  Week 12 | 69.3 | 19.9
  Week 16 (Primary Endpoint) | 78.1 | 18.4

2. Secondary Outcome: Upper Eyelash Length as Measured by Digital Image Analysis in Terms of Change From Baseline to Week 16
Description: Upper eyelash length technologically measured in millimeters
Time Frame: Baseline to Week 16
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
millimeters
  Day 1 (Baseline) | 5.79 (0.815) | 5.71 (0.814)
  Week 1 | 0.05 (0.327) | 0.00 (0.327)
  Week 4 | 0.22 (0.371) | 0.06 (0.382)
  Week 8 | 0.64 (0.559) | 0.07 (0.396)
  Week 12 | 1.16 (0.722) | 0.05 (0.425)
  Week 16 (Primary Endpoint) | 1.39 (0.908) | 0.11 (0.425)

3. Secondary Outcome: Upper Eyelash Length as Measured by Digital Image Analysis in Terms of Change From Baseline to Week 20 (Post-treatment)
Description: Upper eyelash length technologically measured in millimeters
Time Frame: Baseline to Week 20
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
millimeters | 1.47 (0.831) | 0.06 (0.431)

4. Secondary Outcome: Upper Eyelash Thickness as Measured by Digital Image Analysis in Terms of Change From Baseline to Week 16
Description: Progressive thickness technologically measured within preset areas of lashes, expressed in pixels as percentage of the area of interest (AOI). 1 pixel is approximately equal to 0.0273 to 0.0274 mm.
Time Frame: Baseline to Week 16
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: percentage of AOI (in pixels)
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
percentage of AOI (in pixels)
  Day 1 (Baseline) | 16.16 (8.089) | 16.66 (7.787)
  Week 1 | 0.94 (3.651) | 0.24 (3.161)
  Week 4 | 1.62 (4.031) | 0.81 (3.639)
  Week 8 | 3.48 (5.148) | 0.75 (4.189)
  Week 12 | 9.30 (7.328) | 0.95 (4.398)
  Week 16 (Primary Endpoint) | 12.21 (8.381) | 1.10 (3.984)

5. Other Pre Specified Outcome: Patient Reported Outcome: Overall Satisfaction With Eyelashes (Single Item) in Terms of Change From Baseline to Week 16
Description: "Overall, how satisfied are you with your eyelashes?"
  Possible Answers on a 5 point scale as follows:
  1. - Very Satisfied
  2. - Satisfied
  3. - Neutral
  4. - Unsatisfied
  5. - Very Unsatisfied
Time Frame: Baseline to Week 16
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
score on a scale
  Day 1 (Baseline) | 4.18 (0.788) | 4.16 (0.789)
  Week 1 | 0.06 (0.466) | -0.06 (0.550)
  Week 4 | -0.25 (0.829) | -0.35 (0.728)
  Week 8 | -0.90 (1.107) | -0.57 (0.943)
  Week 12 | -1.48 (1.207) | -0.67 (0.939)
  Week 16 (Primary Endpoint) | -1.89 (1.253) | -0.70 (1.074)

6. Primary Outcome: Percentage of Participants Experiencing at Least a 1-grade Increase on the Global Eyelash Assessment (GEA) Scale From Baseline to Week 20 (Post-treatment)
Description: as for outcome 1
Time Frame: Baseline to Week 20
Population: Intent to Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
Percentage of participants | 78.6 | 21.4

7. Secondary Outcome: Upper Eyelash Thickness as Measured by Digital Image Analysis in Terms of Change From Baseline to Week 20 (Post-treatment)
Description: as for outcome 4
Time Frame: Baseline to Week 20
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: percentage of AOI (in pixels)
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
percentage of AOI (in pixels) | 11.16 (7.051) | 1.88 (4.470)

8. Secondary Outcome: Upper Eyelash Darkness as Measured by Digital Image Analysis in Terms of Change From Baseline to Week 16
Description: Darkness was technologically measured in intensity units ranging from 0 (black) - 255 (white)
Time Frame: Baseline to Week 16
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: intensity unit
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
intensity unit
  Day 1 (Baseline) | 105.67 (20.349) | 102.82 (18.161)
  Week 1 | -2.97 (8.102) | -1.25 (8.233)
  Week 4 | -5.10 (10.327) | -2.91 (9.363)
  Week 8 | -9.11 (11.824) | -2.46 (11.249)
  Week 12 | -16.68 (13.585) | -4.22 (11.073)
  Week 16 (Primary Endpoint) | -20.15 (16.051) | -3.57 (10.491)

9. Secondary Outcome: Upper Eyelash Darkness as Measured by Digital Image Analysis in Terms of Change From Baseline to Week 20 (Post-treatment)
Description: Darkness was technologically measured in intensity units ranging from 0 (black) - 255 (white)
Time Frame: Baseline to Week 20
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: intensity unit
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
intensity unit | -20.12 (14.943) | -5.51 (10.789)

10. Other Pre Specified Outcome: Patient Reported Outcome: Overall Satisfaction With Eyelashes (Single Item) in Terms of Change From Baseline to Week 20 (Post-treatment)
Description: "Overall, how satisfied are you with your eyelashes?" Possible Answers on a 5 point scale as follows: (1 - Very Satisfied; 2 - Satisfied; 3 - Neutral; 4 - Unsatisfied; 5 - Very Unsatisfied)
Time Frame: Baseline to Week 20
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Number analyzed (Participants) | 137 | 141
score on a scale | -2.06 (1.345) | -0.61 (1.128)

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.03% Solution | Vehicle Solution
Serious Adverse Events (participants affected / at risk) | 1 | 2
Other Adverse Events (participants affected / at risk) | 40 | 22
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Bimatoprost 0.03% Solution | Vehicle Solution
Squamous cell carcinoma of the skin (back) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/137 | 0/141
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/137 | 1/141
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/137 | 1/141
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Bimatoprost 0.03% Solution | Vehicle Solution
Eye pruritus (Eye disorders) | 5/137 | 1/141
Conjunctival hyperaemia (Eye disorders) | 5/137 | 0/141
Pinguecula (Eye disorders) | 3/137 | 3/141
Eye Irritation (Eye disorders) | 3/137 | 2/141
Dry Eye (Eye disorders) | 3/137 | 1/141
Erythema of eyelid (Eye disorders) | 3/137 | 1/141
Eyelids pruritus (Eye disorders) | 1/137 | 2/141
Conjunctival haemorrhage (Eye disorders) | 0/137 | 2/141
Seasonal allergy (Immune system disorders) | 2/137 | 0/141
Upper respiratory tract infection (Infections and infestations) | 2/137 | 5/141
Sinusitis (Infections and infestations) | 2/137 | 2/141
Influenza (Infections and infestations) | 2/137 | 0/141
Urinary Tract Infection (Infections and infestations) | 1/137 | 2/141
Blepharal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/137 | 0/141
Skin Hyper pigmentation (Skin and subcutaneous tissue disorders) | 4/137 | 1/141
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2/137 | 0/141

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least ninety (90) days prior to any proposed submission for publication or presentation of Study data or other findings related to the Study, the Institution will provide the Sponsor with a manuscript of such submission(s) for review and comment.